CLINICAL TRIAL: NCT01727401
Title: Thromboprophylaxis With Fondaparinux of Deep Vein Thrombosis and Pulmonary Embolism in the Acutely-ill Medical Inpatients With Thrombocytopenia
Brief Title: Thromboprophylaxis of Venous Thromboembolism in Acutely-ill Medical Inpatients With Thrombocytopenia
Acronym: FAITH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Marcello Di Nisio, Principal Investigator, G. d'Annunzio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 213/2012
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Medical Patient; Thrombocytopenia
Keywords: Fondaparinux; medical patient; vein thromboembolism; prophylaxis; thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fondaparinux (Experimental): Drug: fondaparinux once daily sc injections 2.5 mg if renal clearance of creatinine above 50 ml/min once daily sc injections 1.5 mg if renal clearance of creatinine between 20 and 50 ml/min
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux — Fondaparinux once daily sc injections at a dose of 2.5 mg if renal clearance of creatinine above 50 ml/min or Fondaparinux once daily sc injections 1.5 mg if renal clearance of creatinine between 20 and 50 ml/min
  Other Names: Arixtra

SUMMARY:
Fondaparinux is a parenteral anticoagulant drug approved for the prophylaxis of venous thromboembolism in high risk medical patients. A relevant proportion of these patients have renal insufficiency and/or thrombocytopenia which represent independent risk factors for bleeding. The risk of bleeding may be increased when fondaparinux is administered to patients with a reduced renal function and/or low platelet count. A lower dose of fondaparinux, 1.5 mg daily, has been approved for patients with renal insufficiency defined by a creatinine clearance between 20 and 50 mL/min. However, to our knowledge, there are no clinical studies that have specifically evaluated prophylaxis with fondaparinux in acutely-ill medical patients with a moderate to severe thrombocytopenia. The scope of this study is to evaluate the safety of fondaparinux in high risk hospitalized medical patients with a moderate to severe thrombocytopeniada defined by a platelet count between 100,000/uL and 30,000/uL.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years;
* hospitalization in an Internal Medicine Unit and a Barbar score of 4 points or above
* Platelet count between 100,000/uL and 30,000/uL
* written informed consent

Exclusion Criteria:

* Active bleeding or bleeding within the previous 3 months;
* Known bleeding diathesis;
* Active gastroduodenal ulcer;
* Severe renal insufficiency defined by a creatinine clearance below 20 mL/min;
* Ongoing treatment with unfractionated heparin, low-moleculr-weight heparin, fondaparinux, or oral anticoagulants Trattamento in corso con eparina non
* Prophylaxis with unfractionated heparin, low-moleculr-weight heparin, or fondaparinux for more than 48 hours;
* double antiplatelet therapy or acetylsalicylic acid at daily doses above 165 mg;
* planned invasive procedure during the period of thromboprophylaxis;
* Hemoglobin values below 9 g/dL;
* AST or ALT above 2 times the uper limit of normal;
* pregnancy or breast feeding;
* life expectancy lower than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Major bleeding | Participants will be followed for the duration of hospital stay up to two days following hospital discharge, an expected average of 2 weeks
  Major bleeding will be defined as overt bleeding associated with: a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or bleeding that occurs in a critical site: intracranial, intra-spinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal or contributing to death.

SECONDARY OUTCOMES:
Clinically relevant non-major bleeding | Participants will be followed for the duration of hospital stay up to two days following hospital discharge, an expected average of 2 weeks
  clinically relevant non-major bleeding will be defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, unscheduled contact (visit or telephone call) with a physician, (temporary) cessation of study treatment, or associated with discomfort for the patient such as pain, or impairment of activities of daily life.
Minor Bleeding | Participants will be followed for the duration of hospital stay up to two days following hospital discharge, an expected average of 2 weeks
  All bleeding events that cannot be classified as major or clinically relevant non-major
Symptomatic venous thromboembolism | Participants will be followed for the duration of hospital stay up to one month after hospital discharge, an expected average of 5 weeks
  Deep vein thrombosis will be confirmed by compression ultrasonography or venography. Pulmonary embolism will be confirmed by spiral computed tomography or V/Q lung scan

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Di Nisio, PhD, Study Chair — G. d'Annunzio University
Locations (1):
- Marcello Di Nisio, Chieti, Italy